CLINICAL TRIAL: NCT00605189
Title: A Randomized, Controlled Trial Examining Cellular Energetics Related To Various Wound Treatment Therapies
Brief Title: A Trial Examining Cellular Energetics Related to Various Wound Treatment Therapies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study no longer met business objectives
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VACP2005-009
Record Dates: First submitted 2007-12-20; First posted 2008-01-30 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- VAC NPWT (Active Comparator)
  Interventions: Device: Powered Suction Pump (VAC Freedom)
- Gauze-Based NPWT (Active Comparator)
  Interventions: Device: Powered Suction Pump
- Moist Wound Therapy (Active Comparator)
  Interventions: Device: MWT

INTERVENTIONS:
Device: Powered Suction Pump (VAC Freedom) — continuous foam based negative pressure wound therapy
  Other Names: VAC Freedom
  Arms: VAC NPWT
Device: Powered Suction Pump — continuous gauze based negative pressure wound therapy
  Other Names: Gauze-Based Negative Pressure Wound Therapy Device
  Arms: Gauze-Based NPWT
Device: MWT — moist wound therapy
  Arms: Moist Wound Therapy

SUMMARY:
A randomized, controlled pilot study examining how cellular energetics related to various wound treatment therapies in patients with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes
* Subject has a diabetic foot ulcer 5cm squared or greater
* Subject's diabetic foot ulcer is chronic

Exclusion Criteria:

* HgbA1c of 12% or greater
* Presence of cellulitis
* Presence of osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayle M Gordillo, MD, Study Director — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- VAC NPWT: Powered Suction Pump (VAC Freedom): continuous suction, foam based negative pressure wound therapy
- Gauze-Based NPWT: Powered Suction Pump: continuous suction; gauze based negative pressure wound therapy
Period: Overall Study
Arm/Group | VAC NPWT | Gauze-Based NPWT | Moist Wound Therapy
Started | 20 | 21 | 9
Completed | 17 | 19 | 9
Not Completed | 3 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Other | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- VAC NPWT: Powered Suction Pump (VAC Freedom): continuous suction
- Gauze-Based NPWT: Powered Suction Pump: continuous suction
- Total: Total of all reporting groups
Arm/Group | VAC NPWT | Gauze-Based NPWT | Moist Wound Therapy | Total
Number analyzed (Participants) | 20 | 21 | 9 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.8) | 53.9 (8.4) | 56.0 (9.1) | 54.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 10
  Male | 15 | 19 | 6 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 1 | 1 | 0 | 2
  Race/Ethnicity: Asian/Pacific Islander | 0 | 1 | 0 | 1
  Race/Ethnicity: Caucasian | 14 | 11 | 6 | 31
  Race/Ethnicity: Hispanic | 4 | 6 | 3 | 13
  Race/Ethnicity: Other, not specified | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 21 | 9 | 50

OUTCOME MEASURES:

1. Primary Outcome: Compare Energy Charge Between Wound Treatment Therapies
Description: Energy charge is a calculated ratio of the parameters ATP (µg), ADP (µg), and AMP (µg) which are measured with the same unit.
  Energy Charge is calculated as follows:
  Energy Charge = (ATP + (0.5 * ADP)) / (ATP + ADP + AMP)
  Where, ATP = Adenosine triphosphate, ADP = Adenosine diphosphate, AMP = Adenosine monophosphate
Time Frame: Day 0, Day 2, Day 7
Population: Energy charge data was not available for all subjects on the study. Data was only recorded for the subjects listed above.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | VAC NPWT | Gauze-Based NPWT | Moist Wound Therapy
Number analyzed (Participants) | 11 | 8 | 9
Ratio
  Day 0 | 0.4732 (0.0333) | 0.5607 (0.1586) | 0.4873 (0.0310)
  Day 2 | 0.4601 (0.1399) | 0.5535 (0.1377) | 0.4927 (0.0379)
  Day 7 | 0.5289 (0.1395) | 0.5322 (0.1510) | 0.5022 (0.0220)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | VAC NPWT | Gauze-Based NPWT | Moist Wound Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/20 | 1/21 | 2/9
Other Adverse Events (participants affected / at risk) | 12/20 | 9/21 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAC NPWT (N=20) | Gauze-Based NPWT (N=21) | Moist Wound Therapy (N=9)
Osteomyelitis (Infections and infestations) | 2 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Haemaglobin decreased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAC NPWT (N=20) | Gauze-Based NPWT (N=21) | Moist Wound Therapy (N=9)
Skin Maceration (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Panniuculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2
Wound Infection (Infections and infestations) | 2 | 0 | 0
Localised Infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2
Chills (General disorders) | 0 | 0 | 2
Chest Pain (General disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Wound Complication (Injury, poisoning and procedural complications) | 2 | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
International Normalised Ratio Increased (Investigations) | 0 | 0 | 1
Urine Output Decreased (Investigations) | 0 | 0 | 1
Red Cell Distribution Width Increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Shock Hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0 | 0
Wound Drainage (Surgical and medical procedures) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1
Acute Renal Failure (Renal and urinary disorders) | 0 | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days